CLINICAL TRIAL: NCT04846504
Title: Accelerating Implementation of Mindful Mood Balance For Moms
Acronym: MMB4Moms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: HealthPartners Institute (Other); Georgia State University (Other); University of Colorado, Boulder (Other); University of Toronto (Other); Emory University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: U19MH121738 (NIH); 5U19MH121738-02 (NIH)
Record Dates: First submitted 2021-03-23; First posted 2021-04-15 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Perinatal Depression
Keywords: Mindfulness Based Cognitive Therapy; Mindfulness; Perinatal Depression

STUDY DESIGN:
Intervention Model Description: Hybrid type III effectiveness implementation model testing implementation strategies at the individual and OB clinical level. Individual level strategies involve randomizing participants to receive telephonic coaching by professional or peer coach. Clinic level strategies involve randomizing OB clinics to use printed materials and/or electronic medical record prompts to recommend/refer participants to the Mindful Mood Balance for Moms (MMB4M) program or to usual care with no recommendations/referrals to the MMBFM program.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MMBFM program with clinician coach support (Active Comparator): Telephonic coaching provided by licensed mental health professionals to support and encourage participants' engagement in and completion of the 8-session online MMBFM program.
  Interventions: Behavioral: MMBFM program with clinician coach support
- MMBFM program with peer coach support (Active Comparator): Telephonic coaching provided by trained peers with lived experience of perinatal depression to support and encourage participants' engagement in and completion of the 8-session online MMBFM program.
  Interventions: Behavioral: MMBFM program with peer coach support
- Patient facing strategy intervention arm (Active Comparator): Centralized outreach and recruitment of women receiving prenatal care by study team using email, letter, or text, without direct involvement of OB providers.
  Interventions: Behavioral: MMBFM program with clinician coach support; Behavioral: MMBFM program with peer coach support; Behavioral: Patient facing strategy intervention arm
- Patient facing plus clinic facing strategy intervention arm (Active Comparator): OB clinic providers' use of printed recruitment materials and/or electronic medical records prompts to recommend/refer women receiving prenatal care to access the MMBFM program. These clinic facing implementation strategies will be added to the patient facing strategies of centralized outreach and recruitment of women receiving prenatal care by study team using email, letter, or text
  Interventions: Behavioral: MMBFM program with clinician coach support; Behavioral: MMBFM program with peer coach support; Behavioral: Patient facing plus clinic facing strategy intervention arm

INTERVENTIONS:
Behavioral: MMBFM program with clinician coach support — Clinician-delivered telephonic coaching to support participants in the Mindful Mood Balance for Moms online course for prevention of depression relapse/recurrence among perinatal women who have had prior episodes of depression but are not currently depressed.
  Arms: MMBFM program with clinician coach support; Patient facing plus clinic facing strategy intervention arm; Patient facing strategy intervention arm
Behavioral: MMBFM program with peer coach support — Peer-delivered telephonic coaching to support participants in the Mindful Mood Balance for Moms online course for prevention of depression relapse/recurrence among perinatal women who have had prior episodes of depression but are not currently depressed. Peers will be women with lived experience of perinatal depression who are trained on the coaching protocol.
  Arms: MMBFM program with peer coach support; Patient facing plus clinic facing strategy intervention arm; Patient facing strategy intervention arm
Behavioral: Patient facing strategy intervention arm — Direct outreach and recruitment of participants into Mindful Mood Balance for Moms study by study teams. Participants will be women receiving prenatal care at the 4 study sites: Kaiser Permanente Colorado, Southern California, and Georgia, and HealthPartners.
  Arms: Patient facing strategy intervention arm
Behavioral: Patient facing plus clinic facing strategy intervention arm — Direct outreach and recruitment of participants into Mindful Mood Balance for Moms study by study teams, plus recommendation of / referral to the Mindful Mood Balance for Moms study by OB clinicians at the 4 study sites. OB clinicians will choose from printed materials (e.g., flyers, posters in exam rooms and waiting rooms, prescription pads) and electronic medical record prompts (e.g., smart lists, dot phrases) to facilitate engagement in the Mindful Mood Balance for Moms course. Participants will be women receiving prenatal care at the 4 study sites: Kaiser Permanente Colorado, Southern California, and Georgia, and HealthPartners.
  Arms: Patient facing plus clinic facing strategy intervention arm

SUMMARY:
The Mindful Mood Balance for Moms (MMBFM) study examines whether using an internet program called Mindful Mood Balance for Moms to deliver Mindfulness Based Cognitive Therapy (MBCT) over an 8-week time period, is effective for reducing depression symptoms among pregnant women with a history of prior depression, and studies the effects of implementation strategies on the reach of the MMBFM program. This study will enroll 470 women from Kaiser Permanente Colorado, Southern California, Georgia.

The investigators will compare clinical outcomes between those that receive mental health clinician coaching and those that receive peer coaching throughout the 8-week program. Survey data will be collected at 4 time points throughout the study (baseline, 12 weeks, 3rd trimester, and 3 months postpartum). The cost-effectiveness of both the clinical and peer coaching models at each health care system will be evaluated.

For the implementation portion of the study, 30 OB clinics across the 4 health systems will be randomized in equal numbers to provide clinician facing implementation strategies (e.g., recruitment flyers, script pads, electronic medical record prompts) to encourage engagement in the MMBFM program or to usual care where women are only recruited by the study team with no clinician involvement. The primary outcome for testing clinician facing implementation strategies is reach, the percentage of women outreached who initially engage in the MMBFM program.

DETAILED DESCRIPTION:
Specific Aims

Informed by the Consolidated Framework for Implementation Research, a leading implementation science framework, this hybrid type III effectiveness implementation study will evaluate specific implementation strategies for MMBFM. Consistent with a hybrid type III study, there are two goals: (1) compare the clinical effectiveness of MMBFM supported by mental health clinician vs. peer coaches in a randomized trial of 470 pregnant women; and (2) compare the reach of MMBFM across OB clinics for two sets of implementation strategies to facilitate access to and initial engagement in MMBFM: patient facing strategies (PFS - direct outreach to women following prenatal visits via secure patient portal, email, text, or mail) vs. patient facing strategies combined with clinician facing strategies (PFS+CFS - Electronic Medical Record (EMR)-embedded prompts for OB providers, printed prescription pads for providers, flyers). A cluster randomized design will be used, randomizing 30 OB clinics across 4 health systems to either of these two implementation conditions, to assess their impact on reach. The investigators will address the following specific aims:

Aim 1: Compare the clinical effectiveness (i.e. engagement and symptom reduction) of MMBFM supported by clinician vs. peer coaches among women with a history of prior depressive episodes. Hypothesis 1: Coaching delivered by mental health clinicians vs. peers with lived experience will be associated with equivalent reductions in depressive symptoms at 6 months post-randomization.

Aim 2: Examine specific mechanisms of action for MMBFM participants receiving clinician vs. peer coaching. Hypothesis 2a: MMBFM participants receiving peer coaching will report less self-stigma and social isolation than those receiving clinician coaching, and MMBFM participants receiving clinician coaching will report less ruminative response to negative affect and greater decentering at 6 months post-randomization than those receiving peer coaching. Hypothesis 2b: Any difference between peer and clinician coaching in depression outcomes will be mediated by treatment-specific targets - at least partially via increased engagement.

Aim 3: Examine the effects of specific implementation strategies on reach of the MMBFM program. Hypothesis 3: Clinician facing implementation strategies (CFS) in combination with patient facing strategies (PFS) will lead to higher rates of reach than patient facing strategies alone.

Aim 4: Estimate the cost-effectiveness of MMBFM supported by clinician vs. peer coaches. Hypothesis 4: MMBFM will be more cost-effective when supported by peer vs. clinician coaches.

The trials of implementation strategies at the individual and clinic levels will be conducted at four health systems representing diversity in geographic location and in racial and ethnic membership: Kaiser Permanente Colorado, Southern California, and Georgia, and HealthPartners in Minnesota. These sites include 95 clinics and more than 400 obstetric clinicians (OB physicians, nurse practitioners, midwives, nurses), providing prenatal care for 53,000 women annually. The implementation trial for Aims 1 and 2 will recruit 470 women following prenatal care visits total across the four health systems and randomize them in equal numbers to participate in one of the two coaching arms for the MMBFM program, lasting 8 weeks. The clinic-level implementation trial (Aim 3) will involve a cluster randomized design in which 30 OB clinics will be recruited from the four health systems and randomized in equal numbers to either the PFS or PFS+CFS intervention arms, lasting 6 months. The individual- and clinic-level trials will be conducted in parallel.

The 8-session MMBFM program teaches mindfulness practice and cognitive behavioral skills to help reduce automatic, depressogenic modes of thoughts, emotions, and sensations. MMBFM is delivered in a mobile first digital format, accessible from desktop or mobile devices, and provided in an individually tailored manner that includes experiential practice, video-based vicarious learning, and didactic information.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older, receiving prenatal care at one of the 4 participating health systems
* 12-24 weeks gestation
* >= 1 prior episode of major depressive disorder, self-reported
* Current Patient Health Questionnaire 9-item (PHQ9) depression score <=9.
* Have internet access through home computer, smart phone, or similar device

Exclusion Criteria:

* Non-English speaking
* Past history of a psychotic, bipolar disorder, or substance misuse disorder within the past 6 months
* Immediate risk of self-harm
* PHQ9 score <5 or >9
* Patients who are on the "do not call" list for research

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 423 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire 9-item (PHQ-9) scores from baseline through 3 months postpartum | Baseline, 3 months post-randomization, 3rd trimester, 3 months postpartum
  Depression symptom severity, scores range from 0 (low) to 27 (high)
Reach | 6 months post-intervention involving patient facing vs. clinician facing implementation strategies
  The percentage of participants who initially engage in the Mindful Mood Balance for Moms course.

SECONDARY OUTCOMES:
Change in Generalized Anxiety Disorder 7-item (GAD-7) questionnaire scores from baseline through 3 months postpartum | Baseline, 3 months post-randomization, 3rd trimester, 3 months postpartum
  Anxiety symptom severity, scores range from 0 (low) to 21 (high)
Change in Perceived Stress Scale scores from baseline through 3 months postpartum | Baseline, 3 months post-randomization, 3rd trimester, 3 months post partum
  Stress symptoms measured by a 10-item likert-type scores range from 0 to 40 with higher scores indicating higher perceived stress.
Change in Attitudes Toward Motherhood (AToM) Scale scores from baseline through 3 months postpartum | Baseline, 3 months post-randomization, 3rd trimester, 3 months post partum
  Change in attitudes toward motherhood. The 12-item AToM will measure participants' attitudes toward their infants using likert-type responses. Scores range from 0 (positive attitudes) to 60 (negative attitudes).
Change in Short Form 12 (SF-12) scores from baseline through 3 months postpartum | Baseline, 3 months post-randomization, 3rd trimester, 3 months post partum
  The SF-12 is a 12-item measure of physical and mental functional status. Scores range from 0 (low functional status) to 100 (high functional status)
The TWente Engagement with Ehealth Technologies Scale (TWEETS) | 3 months post-randomization
  TWEETS will measure user engagement with the Mindful Mood Balance for Moms program. TWEETS is a 9-item Likert-type scale with scores ranging from 9 (high engagement) to 45 (low engagement)
Client Satisfaction Questionnaire (CSQ) | 3 months post-randomization
  The CSQ will measure satisfaction with the Mindful Mood Balance for Moms program. It is an 8-item questionnaire using different Likert-type responses for each item. Scores range from 8 to 32, with higher values indicating higher satisfaction.

OTHER OUTCOMES:
Change in Ruminative Responses Scale (RRS) short form scores from baseline through 3 months post-randomization | Baseline, 3 months post-randomization
  The 10-item RRS will measure rumination in response to negative affect using likert-type items. Scores range from 10 (low rumination) to 40 (high rumination)
Change in Experiences Questionnaire (EQ) scores from baseline through 3 months post-randomization | Baseline, 3 months post-randomization
  The EQ is a 20-item likert-type scale measuring participant's abilities to decenter, i.e., the ability of viewing the self as separate and different from its own thoughts, the capacity of non-reacting to negative experiences, as well as the ability to be self-compassionate. scores range from 20 (low decentering) to 80 (high decentering).
Change in University of California, Los Angeles (UCLA) Loneliness Scale (ULS-6) scores scores from baseline through 3 months post-randomization | Baseline, 3 months post-randomization
  The ULS-6 is a 6-item scale measuring social isolation using likert-type items. Scores range from 0 (low social isolation) to 18 (high social isolation).
Change in Self-stigma of depression scale (SSDS) scores scores from baseline through 3 months post-randomization | Baseline, 3 months post-randomization
  The SSDS is a 16-item likert-type scale measuring one's perceived self-stigma with depression. Scores range from 16 (high self-stigma) to 80 (low self-stigma).
Attitudes toward coaches | Baseline
  Participants' ratings of their level of comfort with clinician and peer coaches using a Likert-type scale for each type of coach, ranging from 1 (not at all comfortable) to 4 (very comfortable)

CONTACTS AND LOCATIONS:
Overall Officials: Arne Beck, PhD, Principal Investigator — Kaiser Permanente
Locations (4):
- United States (4):
  - Kaiser Permanente Southern California, San Diego, California
  - Kaiser Permanente Colorado, Denver, Colorado
  - Kaiser Permanente Georgia, Atlanta, Georgia
  - HealthPartners, Bloomington, Minnesota

IPD SHARING:
Plan to Share IPD: No